CLINICAL TRIAL: NCT04987788
Title: e-Motivación: Developing and Pilot Testing an App to Improve Latinos' Screening Colonoscopy Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Department of Health and Human Services (U.S. Federal Agency); University of Virginia (Other)
Responsible Party: Principal Investigator, Sarah Miller, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY-18-00328-MOD003; R34AG059705 (NIH)
Record Dates: First submitted 2021-07-23; First posted 2021-08-03 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
Keywords: Colonoscopy; Early Detection of Cancer; Cancer Screening Tests; Motivational Interviewing; Mobile Health; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motívate group (Experimental): Participants will engage with an app on an iPad, smartphone or computer.
  Interventions: Behavioral: Motívate
- Control Group (Active Comparator): Participant receive a link to watch a general health information video.
  Interventions: Behavioral: Video link

INTERVENTIONS:
Behavioral: Motívate — The Motívate app can be used in English or Spanish and involves four sequential phases. 1) The engaging phase uses videos to welcome participants. 2) Patients willing to discuss the decision to have a screening colonoscopy will answer multiple-choice questions on colorectal cancer prevention - completing the focusing phase. Optional videos will offer additional information. 3) The evoking phase consists of interactive Motivational Interviewing exercises to help participants elicit motivations to get a screening colonoscopy. 4) During the planning phase, participants will view a video that will discuss the steps needed to prepare for the colonoscopy.
  Arms: Motívate group
Behavioral: Video link — General health information video link
  Arms: Control Group

SUMMARY:
Among Latinos, a fast growing and underserved population, Colorectal Cancer (CRC) is the third leading cause of cancer death in men and in women. Compared to non-Latino whites, Latinos are less likely to be diagnosed with localized CRC and more likely to be diagnosed with advanced stage disease. Of the recommended CRC screening tests, a colonoscopy allows for both the detection and removal of precancerous and cancerous polyps. Although screening colonoscopies can detect and prevent CRC, more than half of Latinos have not received a screening colonoscopy within the recommended time frame (one screening colonoscopy per ten years).

The purpose of this study is to develop and begin to test an electronically-delivered motivational interviewing progressive web application (e-MI app), called Motívate. The Motívate app will be offered in both English and Spanish to patients who self-identify as Latino/a/x, after they receive a referral for a screening colonoscopy.

DETAILED DESCRIPTION:
A pilot study will be conducted to begin to examine the efficacy of the Motívate app for improving screening colonoscopy uptake among Latinos. Participants (N=80) will be randomly assigned, stratified for language, to one of two groups: Motívate app (N=40) or general health information video (N=40). The results of the pilot study will inform power calculations for a future randomized clinical trial that will formally test the efficacy of the app. If this program of research proves the Motívate app efficacious there is a strong argument to integrate the app into standard clinical care in order to reduce the overall burden of CRC in the growing and vulnerable Latino community.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Latino/a/x;
* English or Spanish-speaking;
* Received a physician referral for a screening colonoscopy;
* Has access to a tablet, smartphone, or computer with working Internet.

Exclusion Criteria:

* Hearing or vision impaired;
* Aim 1 or 2 participant.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J. Miller, PsyD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Proposals should be directed to sarah.miller@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Upon request, we will provide the de-identified dataset to qualified investigators under a Data Use Agreement that provides for: 1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology; and, (3) a commitment to destroying or returning the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motívate Group | Control Group
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motívate Group | Control Group | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (8.14) | 52.9 (5.82) | 53.2 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 20 | 42
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 9 | 4 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Colonoscopy Completion
Description: Screening colonoscopy completion status in medical charts six months after participants are enrolled in the study.
Time Frame: Six months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Motívate Group | Control Group
Number analyzed (Participants) | 22 | 20
Participants | 19 | 19

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Motívate Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT04987788/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT04987788/ICF_001.pdf